CLINICAL TRIAL: NCT00025610
Title: European Infant Neuroblastoma Study - Stage 4S and Stage 4 (No Bone, Lung, Pleura or CNS); MYCN Not Amplified
Brief Title: Combination Chemotherapy in Treating Infants With Newly Diagnosed Neuroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Infant Neuroblastoma Study Group - 1999 (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068979; EURO-INF-NB-STUDY-1999-99.2; EU-20125B
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2001-11

CONDITIONS: Neuroblastoma
Keywords: disseminated neuroblastoma; stage 4S neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Carboplatin; Cyclophosphamide; Doxorubicin; Etoposide; Vincristine

INTERVENTIONS:
Drug: carboplatin
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of different combination chemotherapy regimens in treating infants who have newly diagnosed neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Confirm that the outcome for infants with newly diagnosed stage IV or IVS neuroblastoma without MYCN amplification is not altered by treatment with etoposide and carboplatin followed by cyclophosphamide, doxorubicin, and vincristine.
* Determine whether deletion of chromosome 1p or diploidy/tetraploidy are prognostic factors in these patients.
* Determine whether there are other prognostic criteria that could be used in future therapeutic stratification of these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to age (under 1 month vs over 1 month).

Infants less than 1 month of age are further stratified according to Philadelphia score (less than 1 vs at least 1). Infants over 1 month of age are also further stratified according to Philadelphia score (less than 2 vs at least 2).

Infants under 1 month of age with Philadelphia score of less than 1 and infants over 1 month of age with Philadelphia score of less than 2 undergo observation only. Infants under 1 month of age with Philadelphia score of at least 1 and infants over 1 month of age with Philadelphia score of at least 2 receive VP-CARBO chemotherapy.

* VP-CARBO chemotherapy: Patients receive etoposide IV over 2 hours and carboplatin IV over 1 hour on days 1-3. Treatment repeats every 21 days for 2 courses. Patients with no response receive CADO chemotherapy.
* CADO chemotherapy: Patients receive cyclophosphamide IV over 1 hour on days 1-5, doxorubicin IV over 6 hours on days 4 and 5, and vincristine IV on days 1 and 5. Treatment repeats every 21 days for a maximum of 4 courses.

Patients are followed within 6 months and then annually for 5 years.

PROJECTED ACCRUAL: A total of 130 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed stage IV or IVS neuroblastoma or ganglioneuroblastoma

  * Metastases confined to marrow, skin, nodes, or liver

    * No metastases to bone (radiologic bone lesions in skeleton), CNS, pleura, or lung
* No MYCN amplification (i.e., fewer than 10 copies)

PATIENT CHARACTERISTICS:

Age:

* Under 12 months at diagnosis

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1999-07; Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary P. Gerrard, MBChB, FRCP, FRCPCH, Study Chair — Children's Hospital - Sheffield
Locations (12):
- St. Anna Children's Hospital, Vienna, Austria
- Universitair Ziekenhuis Gent, Ghent, Belgium
- Rigshospitalet, Copenhagen, Denmark
- Centre Hospitalier Regional de Purpan, Toulouse, France
- Istituto Giannina Gaslini, Genoa, Italy
- Rikshospitalet University Hospital, Oslo, Norway
- Instituto Portugues de Oncologia de Francisco Gentil - Centro Regional de Oncologia de Lisboa, S.A., Lisbon, Portugal
- Hospital Universitario LA FE, Valencia, Spain
- Ostra Sjukhuset, Gothenburg, Sweden
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland
- United Kingdom (2):
  - Bristol Royal Hospital for Children, Bristol, England
  - Children's Hospital - Sheffield, Sheffield, England

REFERENCES:
- [Background] De Bernardi B, Gerrard M, Boni L, Rubie H, Canete A, Di Cataldo A, Castel V, Forjaz de Lacerda A, Ladenstein R, Ruud E, Brichard B, Couturier J, Ellershaw C, Munzer C, Bruzzi P, Michon J, Pearson AD. Excellent outcome with reduced treatment for infants with disseminated neuroblastoma without MYCN gene amplification. J Clin Oncol. 2009 Mar 1;27(7):1034-40. doi: 10.1200/JCO.2008.17.5877. Epub 2009 Jan 26. PMID 19171711